CLINICAL TRIAL: NCT07013110
Title: An Artificial Intelligence-powered Approach to Precision Immunotherapy of Human Arthritis - A Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: An Artificial Intelligence-powered Approach to Precision Immunotherapy of Human Arthritis
Acronym: dnaJP1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prof Salvatore Albani (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor-Investigator, Prof Salvatore Albani, Director, SingHealth Translational Immunology and Inflammation Centre (STIIC), Singapore Health Services
Organization: Singapore Health Services (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: dnaJP1
Record Dates: First submitted 2025-05-07; First posted 2025-06-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis (RA); Rheumatology
Keywords: Rheumatoid Arthritis; Rheumatology; dnaJP1; Immune Tolerance
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- dnaJP1 (Experimental): dnaJP1 peptide 25mg with Hydroxychloroquine (HCQ) 200mg once daily are administered orally, preferably in the morning on an empty stomach.
  Interventions: Drug: dnaJP1
- Control (Placebo Comparator): Placebo 25mg with Hydroxychloroquine (HCQ) 200mg once daily are administered orally, preferably in the morning on an empty stomach.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dnaJP1 — The study drug is dnaJP1 peptide. It is a manmade short protein that can be taken easily as a pill. dnaJP1 works to restore the body's immune tolerance by improving its ability to self-adjust - helps to restore the immune system and improve controls on inflammation that has been lost.
  Arms: dnaJP1
Drug: Placebo — This is the control.
  Arms: Control

SUMMARY:
This clinical study is a multi-center, randomized, double-blind, placebo-controlled, outpatient study comparing the efficacy of combination of dnaJP1 peptide and hydroxychloroquine versus combination of placebo and hydroxychloroquine in patients with moderately to severely active RA who are naive to cs-, b-, tsp.-DMARDs.

A sample size of 124 patients will be enrolled in the study. Each patient will receive either combination of dnaJP1 peptide and hydroxychloroquine or combination of placebo and hydroxychloroquine in 1:1 allocation ratio.

DETAILED DESCRIPTION:
Despite the availability of a plethora of new drugs to treat Rheumatoid Arthritis (RA), a holistic and accurate understanding of how therapy with biologics works is still missing. The knowledge gap is particularly poignant if one considers that the second-generation drugs developed for immune therapy is still entirely suppressive. Thus, the dramatic advances in molecular immunology has yet to be translated into the needed evolution from immune suppression to true immune tolerization, an important step on the evolutionary pathway from therapy to cure.

This study is designed to be a multi-center, randomized, double-blind, placebo-controlled trial which has two fundamental objectives:

To identify and dissect mechanisms of induction of immune tolerance in RA patients in response to immune therapy with dnaJP1, a microbiome-derived peptide. Tangibly in the context of clinical development, the investigators aim to capitalize on this knowledge to identify and validate biomarkers predictor of efficacy and clinical response;

The investigators will also determine the effect size needed to demonstrate whether the combination of dnaJP1 peptide and hydroxychloroquine (HCQ) is superior to the combination of placebo and hydroxychloroquine in the treatment of patients with moderately to severely active RA naïve to disease modifying anti-rheumatic drugs (i.e. DMARDs and biologics-naïve).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of rheumatoid arthritis (RA) based on 2010 ACR/EULAR classification criteria
2. DAS28-ESR score more than 3.2 (at least moderately active)
3. Male or female with age 21 or above
4. Ability to understand and sign informed consent
5. Agree to use acceptable methods of contraception for e.g. oral contraceptive pills, implanted contraception, barrier methods, and intra-uterine devices
6. Allowed used of oral Prednisone up to 10 mg/day and NSAIDs, as prescribed by the treating physician
7. Able and willing to comply with the protocol, including availability for all scheduled study visits and assessments.

Using the 2010 ACR/EULAR classification criteria for RA, classification as definite RA is based upon the presence of synovitis in at least one joint, the absence of an alternative diagnosis that better explains the synovitis, and the achievement of a total score of at least 6 (of a possible 10) from the individual scores in four domains. The highest score achieved in a given domain is used for this calculation. These domains and their values are:

1. Number and site of involved joints:

   * 2 to 10 large joints (from among shoulders, elbows, hips, knees, and ankles) = 1 point
   * 1 to 3 small joints (from among the metacarpophalangeal joints, proximal interphalangeal joints, second through fifth metatarsophalangeal joints, thumb interphalangeal joints, and wrists) = 2 points
   * 4 to 10 small joints = 3 points
   * Greater than 10 joints (including at least 1 small joint) = 5 points
2. Serological abnormality (rheumatoid factor or anti-citrullinated peptide/protein antibody)

   * Low positive (above the upper limit of normal [ULN]) = 2 points
   * High positive (greater than three times the ULN) = 3 points
3. Elevated acute phase response (erythrocyte sedimentation rate [ESR] or C-reactive protein [CRP]) above the ULN = 1 point
4. Symptom duration at least six weeks = 1 point

Exclusion Criteria:

1. On prednisolone >10 mg daily
2. History of receiving:

   * conventional synthetic (cs-) disease modifying anti-rheumatic drugs (DMARDs) such as sulfasalazine, methotrexate, and leflunomide administered 6 months prior to screening

     •. biological (b-) DMARDs such as rituximab, infliximab, tocilizumab, adalimumab, etc.
   * tissue-specific (tsp.-) DMARDs such as JAK inhibitors
3. History of lymphoma
4. Active malignancy requiring treatment the last 5 years except for non-melanoma skin cancers and carcinoma of the cervix in situ
5. Pregnancy
6. Breast-feeding
7. Active Infection, e.g., Hepatitis B, tuberculosis
8. A known hypersensitivity to dnaJP1 or to any of the excipients
9. Significant cardiac history, e.g., have experienced any of the following within 12 weeks of study entry: myocardial infarction, unstable ischemic heart disease, stroke, or New York Heart Association Stage IV heart failure
10. A history or presence of dermatological, cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, haematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute a risk when taking HCQ and/or the investigational product or could interfere with the interpretation of data
11. An eGFR based on the most recent available serum creatinine using the Modification of Diet in Renal Disease (MDRD) method of <40 ml/min/1.73 m2
12. A history of chronic liver disease with the most recent available aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the ULN or the most recent available total bilirubin 1.5 times the ULN

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
To estimate effect size needed to ascertain the power i.e. the number of patients to be tested in the future study to prove superiority of the combination dnaJP1 and HCQ versus placebo and HCQ - To determine this ACR20 will be employed | At Study End being 7 Months
  An American College of Rheumatology (ACR) 20% response (ACR20) response was defined as at least 20% improvement in both the tender joint count and the swollen joint count and at least 20% improvement in 3 of the 5 other core set measures listed below.
  The core set required the inclusion of 7 clinical end points for all RA trials: swollen joint count, tender joint count, physician's assessment of disease activity, patient's assessment of disease activity, patient's assessment of pain, and patient's assessment of physical function, and levels of an acute-phase reactant (either the C-reactive protein [CRP] level or the erythrocyte sedimentation rate [ESR]).
A primary endpoint of the study will be to determine safety and tolerability of the experimental treatment in terms of AEs, SAEs, TEAEs | At Study End being 7 Months
  Reporting of Adverse Events
A mechanistic predictor of clinical efficacy at enrolment before first dosing related to immune changes in the cell activation | At Study End being 7 Months
  A combination of high dimensionality technologies will be employed, which will include single cell proteomics, a single cell RNA SEQ flow cytometry and mechanistic studies in vitro
A mechanistic biomarker of treatment response based on 20% change from baseline in increase in Tregs and decrease in inflammatory T cells | At Study End being 7 Months
  Immunological analysis performed on patients samples

SECONDARY OUTCOMES:
To estimate the effect size needed to ascertain the power i.e. the number of patients to be tested in the future study to prove superiority of the combination dnaJP1 and HCQ versus placebo and HCQ - ACR50 | At Study End being 7 Months
  The American College of Rheumatology (ACR) 50% response (ACR50) response is the same instruments with improvement levels defined as 50% versus 20% for ACR20
To estimate the effect size needed to ascertain the power i.e. the number of patients to be tested in the future study to prove superiority of the combination dnaJP1 and HCQ versus placebo and HCQ - ACR70 | At Study End being 7 Months
  The American College of Rheumatology (ACR) 70% response (ACR70) response is the same instruments with improvement levels defined as 70% versus 20% for ACR20
To estimate the effect size needed to ascertain the power i.e. the number of patients to be tested in the future study to prove superiority of the combination dnaJP1 and HCQ versus placebo and HCQ - DAS28-ESR | At Study End being 7 Months
  Disease Activity Score-28 for Rheumatoid Arthritis with erythrocyte sedimentation rate (DAS28- ESR) describes severity of rheumatoid arthritis using clinical and laboratory data, specifically ESR. The number "28" describes the number of different joints examined in the assessment. The DAS-ESR values range from 2.0 to 10.0 while higher values indicate higher disease activity.
  A DAS28-ESR score of ≤ 2.6 indicates remission or ≤ 3.2 indicates low disease activity.
To estimate the effect size needed to ascertain the power i.e. the number of patients to be tested in the future study to prove superiority of the combination dnaJP1 and HCQ versus placebo and HCQ - DAS28-hsCRP | At Study End being 7 Months
  Disease Activity Score-28 for Rheumatoid Arthritis with CRP (DAS28-CRP) is a modification of the DAS28-ESR, DAS28-CRP uses the C-Reactive Protein (CRP) value instead of erythrocyte sedimentation rate (ESR). The DAS28-CRP values range from 2.0 to 10.0 while higher values indicate higher disease activity.
To estimate the effect size needed to ascertain the power i.e. the number of patients to be tested in the future study to prove superiority of the combination dnaJP1 and HCQ versus placebo and HCQ - Clinical Disease Activity Index (CDAI) Score | At Study End being 7 Months
  The CDAI is a composite index (without acute-phase reactant) for assessing disease activity. CDAI score is based on the simple summation of the count of swollen/tender joint count of 28 joints along with patient and physician global assessment on VAS (0-10 cm) Scale for estimating disease activity. The CDAI score ranges from 0 to 76. A CDAI score of ≤ 2.8 indicates remission of disease.
To estimate the effect size needed to ascertain the power i.e. the number of patients to be tested in the future study to prove superiority of the combination dnaJP1 and HCQ versus placebo and HCQ - Simplified Disease Activity Index (SDAI) | At Study End being 7 Months
  The SDAI is the numerical sum of five outcome parameters: tender and swollen joint count (based on a 28-joint assessment), patient and physician global assessment of disease activity [visual analogue scale (VAS) 0-10 cm] and level of C-reactive protein (mg/dl, normal <1 mg/dl). A SDAI score of ≤ 3.3 indicates remission of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Albani, MD PhD, Principal Investigator — Singapore Health Services
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No